CLINICAL TRIAL: NCT04198012
Title: An Open Label Study to Allow Patients Continuous Use of the HemoCare™ Hemodialysis System for Home Hemodialysis Prior to Market Authorization
Brief Title: An Open Label Study to Allow Patients Continuous Use of the HemoCare™ Hemodialysis System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deka Research and Development (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DKPL-00674-001
Record Dates: First submitted 2019-12-05; First posted 2019-12-13 (Actual); Results first posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: End Stage Renal Disease
Keywords: HemoCare™ Hemodialysis System; HemoCare™; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This is an open-label rollover study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- The HemoCare™ Hemodialysis System (Experimental): The HemoCare™ Hemodialysis System is intended for hemodialysis treatment, including short daily and nocturnal hemodialysis, of renal failure patients. The HemoCare™ Hemodialysis System is intended for use in chronic dialysis facilities, self-care dialysis facilities, or the home setting. All treatments must be prescribed by a physician and administered by a trained operator. Treatments must be performed under the supervision or assistance of a medical professional or a care partner who has been trained and deemed competent in the use of the device by the prescribing physician.
  Interventions: Device: HemoCare™ Hemodialysis System

INTERVENTIONS:
Device: HemoCare™ Hemodialysis System — The HemoCare™ Hemodialysis System is intended for hemodialysis treatment, including short daily and nocturnal hemodialysis, of renal failure patients. The HemoCare™ Hemodialysis System is intended for use in chronic dialysis facilities, self-care dialysis facilities, or the home setting. All treatments must be prescribed by a physician and administered by a trained operator. Treatments must be performed under the supervision or assistance of a medical professional or a care partner who has been trained and deemed competent in the use of the device by the prescribing physician.

SUMMARY:
This study is designed to monitor and assess the safety of continued access to the HemoCare™ Hemodialysis System used during the review of the pre-market notifications for the devices in the HemoCare™ Hemodialysis System.

ELIGIBILITY:
Inclusion Criteria:

* Completed DEKA Protocol DKPL 00057 001 and are qualified to enter the study based on the assessment of the Investigator.
* Are willing to comply and capable of complying with the study requirements for therapy with the HemoCare™ Hemodialysis System.
* Have a trained study care partner able to support subject for all at-home study treatments.
* Subject and care partner can read and understand English and provide written informed consent.
* Have a stable functioning vascular access as judged by the treating physician.

Exclusion Criteria:

* Have a current self-reported pregnancy or are actively planning to become pregnant within the next 12 months, lactating, or not using medically acceptable means of contraception during the study.
* Have any any other clinically significant medical disease or condition or subject responsibility that, in the Investigator's opinion, may interfere with a subject's (and/or care partner's) ability to give informed consent, adhere to the protocol, interfere with assessment of the investigational product (IP), or serve as a contraindication to the subject's participation in the study.
* Have a significant psychiatric disorder or mental disability that could interfere with the subject's ability to provide informed consent and/or comply with study procedures.
* Are participating or planning to participate in any other interventional studies except DKPL-00057-001.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - DCI North Brunswick, North Brunswick, New Jersey
  - The Rogosin Institute, New York, New York
  - Dialysis Clinic, Inc., Knoxville, Tennessee
  - Dialysis Clinic, Inc., Nashville, Tennessee
  - Wellbound South Austin, Austin, Texas
  - Wellbound North Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eloot S, Van Biesen W, Dhondt A, Van de Wynkele H, Glorieux G, Verdonck P, Vanholder R. Impact of hemodialysis duration on the removal of uremic retention solutes. Kidney Int. 2008 Mar;73(6):765-70. doi: 10.1038/sj.ki.5002750. Epub 2007 Dec 26. PMID 18160958
- [Background] Culleton BF, Walsh M, Klarenbach SW, Mortis G, Scott-Douglas N, Quinn RR, Tonelli M, Donnelly S, Friedrich MG, Kumar A, Mahallati H, Hemmelgarn BR, Manns BJ. Effect of frequent nocturnal hemodialysis vs conventional hemodialysis on left ventricular mass and quality of life: a randomized controlled trial. JAMA. 2007 Sep 19;298(11):1291-9. doi: 10.1001/jama.298.11.1291. PMID 17878421
- [Background] Rocco MV, Lockridge RS Jr, Beck GJ, Eggers PW, Gassman JJ, Greene T, Larive B, Chan CT, Chertow GM, Copland M, Hoy CD, Lindsay RM, Levin NW, Ornt DB, Pierratos A, Pipkin MF, Rajagopalan S, Stokes JB, Unruh ML, Star RA, Kliger AS; Frequent Hemodialysis Network (FHN) Trial Group; Kliger A, Eggers P, Briggs J, Hostetter T, Narva A, Star R, Augustine B, Mohr P, Beck G, Fu Z, Gassman J, Greene T, Daugirdas J, Hunsicker L, Larive B, Li M, Mackrell J, Wiggins K, Sherer S, Weiss B, Rajagopalan S, Sanz J, Dellagrottaglie S, Kariisa M, Tran T, West J, Unruh M, Keene R, Schlarb J, Chan C, McGrath-Chong M, Frome R, Higgins H, Ke S, Mandaci O, Owens C, Snell C, Eknoyan G, Appel L, Cheung A, Derse A, Kramer C, Geller N, Grimm R, Henderson L, Prichard S, Roecker E, Rocco M, Miller B, Riley J, Schuessler R, Lockridge R, Pipkin M, Peterson C, Hoy C, Fensterer A, Steigerwald D, Stokes J, Somers D, Hilkin A, Lilli K, Wallace W, Franzwa B, Waterman E, Chan C, McGrath-Chong M, Copland M, Levin A, Sioson L, Cabezon E, Kwan S, Roger D, Lindsay R, Suri R, Champagne J, Bullas R, Garg A, Mazzorato A, Spanner E, Rocco M, Burkart J, Moossavi S, Mauck V, Kaufman T, Pierratos A, Chan W, Regozo K, Kwok S. The effects of frequent nocturnal home hemodialysis: the Frequent Hemodialysis Network Nocturnal Trial. Kidney Int. 2011 Nov;80(10):1080-91. doi: 10.1038/ki.2011.213. Epub 2011 Jul 20. PMID 21775973
- [Background] Pauly RP, Gill JS, Rose CL, Asad RA, Chery A, Pierratos A, Chan CT. Survival among nocturnal home haemodialysis patients compared to kidney transplant recipients. Nephrol Dial Transplant. 2009 Sep;24(9):2915-9. doi: 10.1093/ndt/gfp295. Epub 2009 Jul 7. PMID 19584107
- [Background] Bernardo AA, Marbury TC, McFarlane PA, Pauly RP, Amdahl M, Demers J, Hutchcraft AM, Leypoldt JK, Minkus M, Muller M, Stallard R, Culleton BF. Clinical safety and performance of VIVIA: a novel home hemodialysis system. Nephrol Dial Transplant. 2017 Apr 1;32(4):685-692. doi: 10.1093/ndt/gfw044. PMID 27190336
- [Background] U.S. Renal Data System. USRDS 2017 Annual Data Report: Atlas of End-Stage Renal Disease in the United States. Bethesda, MD: National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases; 2017

RESULTS

PARTICIPANT FLOW:
Groups:
- The HemoCare™ Hemodialysis System: All subjects who complete DEKA Protocol DKPL-00057-001 and meet all of the inclusion criteria and exclusion criteria will.
Period: Overall Study
Arm/Group | The HemoCare™ Hemodialysis System
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | The HemoCare™ Hemodialysis System
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.24 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Safety Event
Description: The Total Number of subjects having at least one Anticipated AE, Unanticipated AE, Device Related AE, Anticipated SAE, Unanticipated SAE and Device Related SAEs.
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | The HemoCare™ Hemodialysis System
Number analyzed (Participants) | 25
participants
  Anticipated Adverse Event | 20
  Unanticipated Adverse Event | 20
  Device-Related Adverse Event | 5
  Anticipated Serious Adverse Event | 6
  Unanticipated Serious Adverse Event | 12
  Device Related Serious Adverse Event | 0

ADVERSE EVENTS:
Time Frame: During study participation - from the time of consent until the end of participation (on average 1 year)
Description: All Adverse Events and Serious Adverse Events were recorded, regardless of relatedness.
Arm/Group | The HemoCare™ Hemodialysis System
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 15/25
Other Adverse Events (participants affected / at risk) | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The HemoCare™ Hemodialysis System (N=25)
Chest discomfort (General disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Arteriovenous fistula site infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 1 (2)
SARS-CoV-2 test positive (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypervolemia (Metabolism and nutrition disorders) | 3 (3)
Bell's palsy (Nervous system disorders) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1)
Renal transplant (Surgical and medical procedures) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The HemoCare™ Hemodialysis System (N=25)
Palpitations (Cardiac disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 2 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 2 (3)
Conjunctivitis (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Localized infection (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 2 (3)
Vascular access site hemorrhage (Injury, poisoning and procedural complications) | 3 (4)
Vascular access site pain (Injury, poisoning and procedural complications) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (4)
Vascular graft complication (Injury, poisoning and procedural complications) | 2 (2)
Blood phosphorus increased (Investigations) | 2 (3)
Blood potassium increased (Investigations) | 2 (2)
Hemoglobin decreased (Investigations) | 4 (5)
Heart rate increased (Investigations) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (9)
Hyperphosphatemia (Metabolism and nutrition disorders) | 3 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (28)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (6)
Metabolic alkalosis (Metabolism and nutrition disorders) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (18)
Dizziness (Nervous system disorders) | 5 (7)
Headache (Nervous system disorders) | 4 (6)
Hypoesthesia (Nervous system disorders) | 2 (2)
Thrombosis in device (Product Issues) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (7)
Hemorrhage (Vascular disorders) | 6 (12)
Hypotension (Vascular disorders) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT04198012/Prot_SAP_001.pdf